CLINICAL TRIAL: NCT03067064
Title: Prevelance of Molar Incisors Hypomineralization Among a Group of Egyptian Children
Brief Title: Prevelance of Molar Incisor Hypomineralization Among a Group of Egyptian Children
Acronym: MIH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Zaki Youssef, master dental student at pediatric dentistry department, Cairo University
Other Study IDs: Ryoussef
Record Dates: First submitted 2017-02-17; First posted 2017-03-01 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Child Development Disorder
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Clinical examination

SUMMARY:
The purpose of this study is to find out the prevalence of molar incisor hypomineralization among a group of Egyptian children

DETAILED DESCRIPTION:
Molar incisor hypomineralization is frequent in many population throughout the world and a wide variation of molar incisior hypomineralization 2.4_40% has been reported.To the best of our knowledge,there is no Sufficient information regarding the prevalence of molar incisor hypomineralization in Egyptian children therefore the aim of this study is to assess the prevalence of molar incisor hypomineralization among a group of Egyptian children.

ELIGIBILITY:
Inclusion Criteria:

- Patient seeks dental care in paediatric dentistry and dental public health department in Cairo university

* positive patient acceptance for participation in the study
* children with at least one of four permanent molars erupted or partially erupted

Exclusion Criteria:

* uncooperative children

  * children with appliance
  * children with systemic diseases

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Group of Egyptian children attending in paediatric dentistry and dental public health department in the faculty of oral and dental medicine,Cairo university
Sampling Method: Probability Sample
Enrollment: 610 (Estimated)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Presence of Molar incisor hypomineralization | 10min
  Presence of Molar incisor hypomineralization or not through clinical examination (binary)

SECONDARY OUTCOMES:
Severity of Molar incisor hypomineralization | 15min
  Clinical examination using modified index based on EAPD criteria

CONTACTS AND LOCATIONS:
Overall Officials: Reem Za Youssef, Bechlor, Principal Investigator — Cairo University
Locations (1):
- Reem Zaki Youssef, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Yannam,s.,Amarlar,D.&Rekha,C.,2016.prevelance of molar incisor hypomineralization in school children aged 8_12years in chennai .journal of indian society of pedodontic and preventive dentistry — http://www.jisppd.com